CLINICAL TRIAL: NCT07098494
Title: Can Probiotics Serve as an Adjuvant Therapy for Post-Pullthrough Hirschsprung's Disease-Associated Enterocolitis?
Brief Title: Probiotics and Post-Pullthrough Hirschsprung's Disease-Associated Enterocolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Magdy Abdelmohsen, Dr., Aswan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AswanUH8
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hirschsprung Disease; Enterocolitis; Hirschsprung's Disease Associated Enterocolitis
Keywords: Hirschsprung disease; enterocolitis; Saccharomyces boulardii; HAEC
MeSH Terms: conditions — Hirschsprung Disease; Enterocolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saccharomyces boulardii probiotics (Experimental)
  Interventions: Dietary Supplement: Saccharomyces Boulardii Probiotic Supplement

INTERVENTIONS:
Dietary Supplement: Saccharomyces Boulardii Probiotic Supplement — • Saccharomyces boulardii (strain CNCM I-745): 250 mg per day (5 billion colony-forming units (CFU)

SUMMARY:
This was a prospective case-controlled study investigating the role of probiotics in the management of Hirschsprung-associated enterocolitis (HAEC). The study was conducted across three children's hospitals in Upper Egypt, spanning from January 2018 to September 2024.

The study was randomized, with parents of the participating children choosing one of two paper forms to become either included in the probiotic treatment regimen or adhere to the standard treatment protocol without probiotics, the latter serving as the control group.

The inclusion criteria encompassed children under 12 years of age and admitted for treatment of a grade II post-pullthrough HAEC episode. Exclusion criteria included patients with severe comorbidities, hemodynamic instability, active septicemia, grade III HAEC, other congenital anomalies, trisomy 21, inability to tolerate or take oral probiotics, probiotic sensitivities, or any contraindications to probiotic use.

DETAILED DESCRIPTION:
This was a prospective case-controlled study investigating the role of probiotics in the management of Hirschsprung-associated enterocolitis (HAEC). The study was conducted across three children's hospitals in Upper Egypt, spanning from January 2018 to September 2024. Diagnosis of Hirschsprung disease (HD) was confirmed through rectal biopsy prior to any surgical intervention. The study was randomized, with parents of the participating children choosing one of two paper forms to become either included in the probiotic treatment regimen or adhere to the standard treatment protocol without probiotics, the latter serving as the control group.

The inclusion criteria encompassed children under 12 years of age and admitted for treatment of a grade II post-pullthrough HAEC episode. Exclusion criteria included patients with severe comorbidities, hemodynamic instability, active septicemia, grade III HAEC, other congenital anomalies, trisomy 21, inability to tolerate or take oral probiotics, probiotic sensitivities, or any contraindications to probiotic use.

Demographic and clinical data were extracted from the medical records, clinical history taken and follow-up, including age, sex, comorbidities, HAEC grade, laboratory parameters, imaging findings, and treatment details. Outcome measures included resolution of HAEC symptoms, duration of hospital stay, recurrence rates, and any complications. Follow-up data were collected for six months following the resolution of acute HAEC symptoms.

The management protocol and medications for standard group

* A clear liquid or nothing by mouth, nasogastric decompression, intravenous fluids calculated by pediatric physician according to the body weight, rectal irrigations once per day.
* Metronidazole 10 mg/kg/dose IV 8 hrs × 10 days, Max. 500 mg/dose. Administer undiluted solution over 20 to 30 minutes.
* Broad spectrum antibiotics as Ampicillin and gentamicin. The pediatrics dose of Ampicillin for children less than 40 kg was 50 mg/kg/day IM or IV in equally divided doses every 8 hours. For children at least 40 kg or more the dose was 500 mg IM or IV every 8 hours. The pediatric dose of gentamicin was 2 to 2.5 mg/kg IM or IV every 8 hours for 7 to 10 days.
* For fever, Perfalgan IV in a dose of 15 mg/kg every 6 hours was useful.
* PPI Omeprazole solution via enteral feeding tubes, in a dose of (1-3mg/kg once daily up to 1-year, max 20mg) (2 - 12 years: 10-19kg, max 20mg) (2 - 12 years: 20kg+, max 40mg).

Probiotic Supplementation for the Probiotics Group:

The probiotic formulation included:

* Saccharomyces boulardii (strain CNCM I-745): 250 mg per day (5 billion colony-forming units (CFU)
* Lactobacillus rhamnosus (strain GG): 5 billion CFU per day
* Bifidobacterium infantis (strain 35624): 5 billion CFU per day
* Administration:

The probiotics were administered in the form of a powder mixed with water or a small amount of clear liquid, ensuring ease of administration for pediatric patients. Probiotic supplementation was administrated once daily in the morning half an hour before any other types of oral feeding. Avoid concurrent antibiotics (space 2 hours apart). It continued for 3 months following the resolution of acute HAEC symptoms.

ELIGIBILITY:
Inclusion Criteria:

* children under 12 years of age
* a grade II post-pullthrough HAEC episode.

Exclusion Criteria:

* patients with severe comorbidities.
* hemodynamic instability.
* active septicemia
* grade III HAEC
* trisomy 21
* inability to tolerate or take oral probiotics
* probiotic sensitivities
* any contraindications to probiotic use.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The clinical outcome as resolution of HAEC symptoms. | 3 MONTHS
  It included the clinical outcome as resolution of HAEC symptoms; defined by improvement of fever, diarrhea, and abdominal distension.

SECONDARY OUTCOMES:
The laboratory outcome | 3 months
  The laboratory outcome as change in the inflammatory markers levels of C-reactive protein (CRP) and white blood cell (WBC) count before and after treatment.
The radiological outcome | 3 months
  The serial changes in the radiological images.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided